CLINICAL TRIAL: NCT03889925
Title: Effect of Different Injection Regimens of Autologous Conditioned Plasma for the Treatment of Symptomatic Knee Osteoarthritis
Brief Title: Effect of Different Injection Regimens of Autologous Conditioned Plasma for Knee Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Andrews Research & Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1379083
Record Dates: First submitted 2019-03-15; First posted 2019-03-26 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid; orthovisc

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the type of injection that they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Autologous conditioned plasma group (Experimental): Participants in this group will receive a three-injection series of autologous conditioned plasma over the course of 3 consecutive weeks.
  Interventions: Biological: Autologous conditioned plasma
- Autologous conditioned plasma with hyaluronic acid group (Experimental): Participants in this group will receive a two-injection series of autologous conditioned plasma and hyaluronic acid (Hymovis, Fidia Pharmaceuticals) and a third injection on the third week of autologous conditioned plasma.
  Interventions: Drug: Hyaluronan

INTERVENTIONS:
Drug: Hyaluronan — Patients will receive 2 intra-articular injections of autologous conditioned plasma and hyaluronic acid once a week for 2 weeks and a third injection on the third week of ACP.
  Other Names: Hymovis; Monovisc; Orthovisc
  Arms: Autologous conditioned plasma with hyaluronic acid group
Biological: Autologous conditioned plasma — Patients will receive 3 intra-articular injections of autologous conditioned plasma dosed at once a week for 3 weeks.
  Arms: Autologous conditioned plasma group

SUMMARY:
The clinical efficacy of hyaluronic acid or corticosteroid injections has been reported, but effects are short lived. This has led to the development of additional injection options such as autologous derived blood products which have been documented to alleviate symptoms related to knee osteoarthritis, with recent comparative studies suggesting a greater, long-lasting effect with these blood derived products like platelet rich plasma (PRP) [2-8]. One clinically-developed preparation of platelet rich plasma, named autologous conditioned plasma (ACP), has randomized controlled trial data proving efficacy [4,9]. Clinical use of platelet rich plasma for knee arthritis typically involves a 3-injection series over 3 weeks, i.e. an injection once a week for three weeks. The main objective of this study is to determine if hyaluronic acid (HA) injected at the same time as autologous conditioned plasma (ACP), a leukocyte-poor platelet rich plasma product, will improve the performance of ACP in the treatment of symptomatic knee osteoarthritis. It is hypothesized that the injection of hyaluronic acid will improve the efficacy of ACP.

DETAILED DESCRIPTION:
Patients between the ages of 30 and 80 who have documented radiographic evidence of OA in the tibiofemoral or patellofemoral compartment of the target knee (Kellgren-Lawrence grades 1-4) will be screened for participation in this study. Patients must have a documented diagnosis of primary OA for at least six weeks. 80 patients will be recruited through the Andrews Institute physician practices. The study design will be a randomized control trial. Participants who meet the inclusion criteria will have the study explained in detail, and informed consent will be obtained as outlined above. Participants will complete patient-reported outcome questionnaires prior to their injection. The questionnaires will include the Western Ontario and McMaster University Osteoarthritis Index (WOMAC), International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC), Knee Injury and Osteoarthritis Outcome Score (KOOS). Participants will also complete these questionnaires at 1, 3, 6, 12, 18, and 24 months after the final injection. A trained medical professional will draw blood from the patient's arm, and the blood will be spun in a centrifuge for 5 minutes at 1500 RPM. The platelets will then be separated for injection into the patient's knee. The treating physician will then inject the ACP into the involved knee joint following standard aseptic technique per the physician's standard of care. This entire process will be completed in a single patient visit. Any unused portion of a sample in the physician's office will be disposed of through standard biohazard waste disposal systems as required by law. Group 1 [ACP]: Will receive three intra-articular injections of autologous conditioned plasma dosed once a week for three weeks. Group 2 [ACP-HA]: Will receive two intra-articular injections of autologous conditioned plasma and hyaluronic acid once a week for two weeks and a third injection on the third week of ACP.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 30 and 80
* Documented radiographic evidence of OA in the tibiofemoral or patellofemoral compartment of the involved knee (Kellgren-Lawrence grades 1-4)
* Patients must have a documented diagnosis of primary OA for at least 6 weeks.

Exclusion Criteria:

* Patients who have had viscosupplementation in the involved knee in the past 6 months.
* Any patient who has had a corticosteroid injection in any joint within 3-months prior to screening will be excluded.
* Patients with gout or rheumatologic disease will be excluded. Patients who have had a previous negative experience with HA.
* Any patient who will have difficulty obtaining internet access, does not have an active e-mail address, or is unable to comprehend study documents or give informed consent will be excluded.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Anz, MD, Principal Investigator — Andrews Institute
Locations (1):
- Andrews Institute for Orthopaedics & Sports Medicine, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spakova T. Re: Treatment of knee joint osteoarthritis with autologous platelet-rich plasma in comparison with hyaluronic acid. Am J Phys Med Rehabil. 2014 Jan;93(1):95. doi: 10.1097/phm.0b013e318282ea04. No abstract available. PMID 24501778
- [Background] Kon E, Mandelbaum B, Buda R, Filardo G, Delcogliano M, Timoncini A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma intra-articular injection versus hyaluronic acid viscosupplementation as treatments for cartilage pathology: from early degeneration to osteoarthritis. Arthroscopy. 2011 Nov;27(11):1490-501. doi: 10.1016/j.arthro.2011.05.011. Epub 2011 Aug 10. PMID 21831567
- [Background] Cerza F, Carni S, Carcangiu A, Di Vavo I, Schiavilla V, Pecora A, De Biasi G, Ciuffreda M. Comparison between hyaluronic acid and platelet-rich plasma, intra-articular infiltration in the treatment of gonarthrosis. Am J Sports Med. 2012 Dec;40(12):2822-7. doi: 10.1177/0363546512461902. Epub 2012 Oct 25. PMID 23104611
- [Background] Patel S, Dhillon MS, Aggarwal S, Marwaha N, Jain A. Treatment with platelet-rich plasma is more effective than placebo for knee osteoarthritis: a prospective, double-blind, randomized trial. Am J Sports Med. 2013 Feb;41(2):356-64. doi: 10.1177/0363546512471299. Epub 2013 Jan 8. PMID 23299850
- [Background] Li M, Zhang C, Ai Z, Yuan T, Feng Y, Jia W. [Therapeutic effectiveness of intra-knee-articular injection of platelet-rich plasma on knee articular cartilage degeneration]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2011 Oct;25(10):1192-6. Chinese. PMID 22069972
- [Background] Filardo G, Kon E, Di Martino A, Di Matteo B, Merli ML, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma vs hyaluronic acid to treat knee degenerative pathology: study design and preliminary results of a randomized controlled trial. BMC Musculoskelet Disord. 2012 Nov 23;13:229. doi: 10.1186/1471-2474-13-229. PMID 23176112
- [Background] Vaquerizo V, Plasencia MA, Arribas I, Seijas R, Padilla S, Orive G, Anitua E. Comparison of intra-articular injections of plasma rich in growth factors (PRGF-Endoret) versus Durolane hyaluronic acid in the treatment of patients with symptomatic osteoarthritis: a randomized controlled trial. Arthroscopy. 2013 Oct;29(10):1635-43. doi: 10.1016/j.arthro.2013.07.264. PMID 24075613
- [Background] Smith PA. Intra-articular Autologous Conditioned Plasma Injections Provide Safe and Efficacious Treatment for Knee Osteoarthritis: An FDA-Sanctioned, Randomized, Double-blind, Placebo-controlled Clinical Trial. Am J Sports Med. 2016 Apr;44(4):884-91. doi: 10.1177/0363546515624678. Epub 2016 Feb 1. PMID 26831629

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autologous Conditioned Plasma Group | Autologous Conditioned Plasma With Hyaluronic Acid Group
Started | 32 | 32
Completed | 21 | 22
Not Completed | 11 | 10
Not completed — Lost to Follow-up | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Conditioned Plasma Group | Autologous Conditioned Plasma With Hyaluronic Acid Group | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.4) | 60.7 (9) | 58.25 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
IKDC [Mean (Standard Deviation); unit: Score] | 39.2 (10.4) | 38.6 (14.5) | 38.9 (12.52)
WOMAC [Mean (Standard Deviation); unit: Score] | 40 (18.6) | 40.5 (18.7) | 40.25 (18.5)
KOOS [Mean (Standard Deviation); unit: Score] | 42.7 (12.7) | 44.3 (14.4) | 43.5 (13.49)

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster University's Osteoarthritis Index (WOMAC)
Description: Patient reported outcome measure; The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of the scores for all three subscales gives a total score. Higher scores indicate worse pain, stiffness, and functional limitations.
Time Frame: Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post injections
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Conditioned Plasma Group | Autologous Conditioned Plasma With Hyaluronic Acid Group
Number analyzed (Participants) | 32 | 32
score on a scale
  1 Month | 24.9 (15.6) | 22.4 (15.2)
  3 Months | 26.1 (20.1) | 22.3 (16.3)
  6 Months | 21.9 (15.3) | 22.5 (16.5)
  12 Months | 25.9 (18.7) | 22.7 (19.3)
  18 Months | 21 (15.1) | 27.1 (23.8)
  24 Months | 26.7 (17.8) | 29.2 (23.3)

2. Primary Outcome: International Knee Documentation Committee Subjective Knee Evaluation Form
Description: Patient reported outcome measure; Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
Time Frame: Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post injections
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Autologous Conditioned Plasma Group | Autologous Conditioned Plasma With Hyaluronic Acid Group
Number analyzed (Participants) | 32 | 32
score on a scale
  1 Month | 50.1 (17.3) | 53.7 (14.1)
  3 Months | 50.4 (17.6) | 56.9 (17.6)
  6 Months | 53.1 (16) | 53.1 (19.9)
  12 Months | 50.6 (19.1) | 55.7 (21.5)
  18 Months | 57 (23.6) | 53.4 (24.5)
  24 Months | 50.9 (20.1) | 51.8 (21.9)

3. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score
Description: Patient reported outcome measure; A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated.
Time Frame: Baseline, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months post injections
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Autologous Conditioned Plasma Group | Autologous Conditioned Plasma With Hyaluronic Acid Group
Number analyzed (Participants) | 32 | 32
score
  1 Month | 59.4 (13.5) | 62.7 (12.5)
  3 Months | 59 (18.8) | 62.9 (20.5)
  6 months | 64.2 (16.3) | 62.5 (18.1)
  12 Months | 61.8 (17.7) | 61.8 (20.4)
  18 Months | 65.3 (18.2) | 59.8 (19.5)
  24 Months | 59.8 (19.5) | 59 (24.4)

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | Autologous Conditioned Plasma Group | Autologous Conditioned Plasma With Hyaluronic Acid Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT03889925/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT03889925/ICF_001.pdf